CLINICAL TRIAL: NCT00991939
Title: Initial Treatment of Patients With Immune Thrombocytopenic Purpura: The ITP^2 Study
Brief Title: Initial Treatment of Patients With Immune Thrombocytopenic Purpura
Acronym: ITP^2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was closed due to accrual futility there were only a total of 8 subjects enrolled.
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 675; U01HL072268 (NIH); HL072268; HL072033; HL072291; HL072196; HL072289; HL072248; HL072191; HL072299; HL072305; HL072274; HL072028; HL072359; HL072072; HL072355; HL072283; HL072346; HL072331; HL072290
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Immune Thrombocytopenic Purpura
Keywords: Immune thrombocytopenic purpura; ITP; Dexamethasone; Prednisone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose pulse dexamethasone (Experimental)
  Interventions: Drug: Dexamethasone USP Micronized
- Standard prednisone therapy (Active Comparator)
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Dexamethasone USP Micronized — The dose for dexamethasone is 30 mg/day for patients < 60 kg and 40 mg/day for patients > 60 kg. The patient will be dosed on days 1-4, 15-18 and 29-32. On the remaining days during the treatment phase of the study, the patient will receive placebo capsules.
  Arms: High dose pulse dexamethasone
Drug: Prednisone — Prednisone will be administered to study patients at a dose of 60 mg/day for patients less than 60 kg and 80 mg/day for patients > 60 kg for 21 days. The following schedule for tapering of prednisone will be used: after three weeks of treatment at either 60 mg/day (for patients < 60 kg) or 80 mg/day (for patients ≥ 60 kg), the dose will be reduced to 40 mg/day for 1 week, then 20 mg/day for 1 week, then 10 mg/day for 1 week, then 5 mg/day for 1 week and then stopped. Placebo capsules will be added as necessary during the treatment phase of the study, to maintain blinding.
  Arms: Standard prednisone therapy

SUMMARY:
This study will compare treatment with 3 courses of high-dose dexamethasone versus treatment with prednisone, for patients recently diagnosed with immune thrombocytopenic purpura (ITP). The primary hypothesis is that patients treated with high-dose dexamethasone will obtain a more durable remission than patients treated with prednisone.

DETAILED DESCRIPTION:
ITP is a common disorder associated with significant morbidity. For more than 40 years it has been recognized that this disorder was responsive to corticosteroid therapy. As corticosteroids are easily obtainable and inexpensive, they have become the standard first-line therapy for adult patients with newly-diagnosed ITP. Generally, patients are treated with prednisone at a dose of approximately 1 mg/kg, or 60 mg/day, and once a response is obtained the daily dosage is gradually tapered. While approximately 70% of patients treated in this manner respond initially, most will relapse as the corticosteroid dose is lowered; ultimately only 15-20% of patients achieve a complete or partial remission of their ITP at an "acceptable" dose of prednisone. Recently, several studies have suggested that the use of high dose corticosteroids, specifically pulse dexamethasone, may be a more efficacious initial therapy for ITP, capable of causing a higher initial response rate and a significantly longer duration of remission despite a shorter course of initial therapy.

This study will compare treatment with 3 courses of high-dose dexamethasone versus treatment with prednisone, for patients recently diagnosed with immune thrombocytopenic purpura (ITP). The primary hypothesis is that patients treated with high-dose dexamethasone will obtain a more durable remission than patients treated with standard oral corticosteroids. This may reflect the ability of high dose corticosteroids to eradicate a sensitive pathogenic lymphoid clone that may be transiently susceptible to aggressive immunosuppressive therapy early in the course of disease.

ELIGIBILITY:
Inclusion Criteria:

* Must meet criteria for a diagnosis of ITP as specified by ASH guidelines
* Must be within 30 days after diagnosis of ITP at the time of randomization (diagnosis of ITP starts with first platelet count ≤ 100,000/μl)
* Platelet count ≤ 30,000/μl at the time ITP is diagnosed, and/or at some time between the diagnosis of ITP and study entry
* Platelet count ≤ 150,000/μl at the time of randomization
* Age ≥ 15 years
* If bone marrow examination is available, it must be compatible with ITP
* Subjects, or their legal guardians, must have the ability to provide informed consent

Exclusion Criteria:

* Rituximab therapy or splenectomy for ITP or for any other cause within the previous 8 weeks.
* Known HIV infection
* Known HCV infection
* Known systemic lupus erythematosus
* Pregnancy or breastfeeding
* Insulin-requiring diabetes mellitus
* Previous exposure to prednisone for ITP at a dose ≥ 1.5 mg/kg prednisone/day for ≥ 1 week prior to study entry
* Ongoing use of treatments that are known to inhibit platelet function, e.g. aspirin
* Anything that in the opinion of the investigator is likely to interfere with participation in the study
* Persons previously randomized in the ITP^2 study
* Persons currently enrolled in other interventional clinical trials
* Exposure to thrombopoietic agent prior to study entry
* Previous exposure to dexamethasone for the treatment of ITP at a dose of 30 mg/day or greater for subjects < 60 kg or 40 mg/day or greater for subjects >= 60 kg for at least four days

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan F Assmann, PhD, Principal Investigator — Carelon Research; James Bussel, MD, Principal Investigator — Weill Medical College, Cornell University; Alvin Schmaier, MD, Principal Investigator — Case Western Reserve University; Jodi Segal, MD, Principal Investigator — Johns Hopkins University; Terry Gernsheimer, MD, Principal Investigator — University of Washington; Eliot Williams, MD, Principal Investigator — University of Wisconsin, Madison; Ellis Neufeld, MD, Principal Investigator — Boston Children's Hospital; Judith Lin, MD, Principal Investigator — Brigham and Women's Hospital; Thomas Ortel, MD, Principal Investigator — Duke University; David Kuter, MD, Principal Investigator — Massachusetts General Hospital; Cindy Leissinger, MD, Principal Investigator — Tulane University; Ann Zimrin, MD, Principal Investigator — University of Maryland; Nigel Key, MD, Principal Investigator — University of North Carolina, Chapel Hill; James George, MD, Principal Investigator — The University of Oklahoma; Michele Lambert, MD, Principal Investigator — Children's Hospital of Philadelphia; Joseph Kiss, MD, Principal Investigator — University of Pittsburgh; Bruce Sachais, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (18):
- United States (18):
  - Tulane University, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - Weill Medical College, Cornell University, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Presbyterian and Shadyside Hospital, Pittsburgh, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
  - Gundersen Clinic, La Crosse, Wisconsin
  - University of Wisconsin, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose Pulse Dexamethasone: Dexamethasone USP Micronized : The dose for dexamethasone is 30 mg/day for patients < 60 kg and 40 mg/day for patients > 60 kg. The patient will be dosed on days 1-4, 15-18 and 29-32. On the remaining days during the treatment phase of the study, the patient will receive placebo capsules.
- Standard Prednisone Therapy: Prednisone : Prednisone will be administered to study patients at a dose of 60 mg/day for patients less than 60 kg and 80 mg/day for patients > 60 kg for 21 days. The following schedule for tapering of prednisone will be used: after three weeks of treatment at either 60 mg/day (for patients < 60 kg) or 80 mg/day (for patients ≥ 60 kg), the dose will be reduced to 40 mg/day for 1 week, then 20 mg/day for 1 week, then 10 mg/day for 1 week, then 5 mg/day for 1 week and then stopped. Placebo capsules will be added as necessary during the treatment phase of the study, to maintain blinding.
Period: Overall Study
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Started | 5 | 3
Completed | 0 | 1
Not Completed | 5 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Entire study terminated | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 1 | 6
  >=65 years | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (15.6) | 62.5 (35.8) | 46.7 (26.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients in Each Treatment Arm Who Remain Free of All ITP Therapy With a Platelet Count ≥ 50,000/μl From 60 Days Through 365 Days After Study Entry.
Time Frame: From 60 days through 365 days after study entry.
Measure: Number; unit: percentage of subjects
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 3 | 1
percentage of subjects | 0 | 0
Statistical Analysis 1: Comparison: High Dose Pulse Dexamethasone vs Standard Prednisone Therapy; Four subjects were not included in this analysis because not enough data was available to assess the primary outcome at the time the study was terminated; Test type: Superiority or Other; p = 1.00, Fisher Exact; Difference of proportions = 0, 95% CI 2-sided [-0.975 to 0.708], Standard Error of Mean 0.58 — The estimated value is the proportion of success in the high dose pulse dexamethasone group minus the proportion of success in the standard prednisone group

2. Secondary Outcome: The Percentage of Patients Who Remain Free of All ITP Therapy With a Platelet Count ≥ 150,000/μl From 60 Days Through 365 Days After Study Entry
Time Frame: From 60 days through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: The Percentage of Patients With Platelets ≥ 50,000/μl at 365 Days Who Are Off All Treatment, Have Received ≤ 2 Acute Therapeutic Interventions for Thrombocytopenia, and Whose Last Acute Therapeutic Intervention Occurred at Least 90 Days Before Day 365
Time Frame: 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: The Percentage of Patients Who Remain Free of All ITP Therapy With a Platelet Count of ≥ 150,000 From 180 Through 365 Days After Study Entry
Time Frame: From 180 days through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: The Percentage of Patients Who Remain Free of All ITP Therapy With a Platelet Count of ≥ 50,000 From 180 Through 365 Days After Study Entry
Time Frame: From 180 days through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: The Percentage of Patients Receiving Acute Therapeutic Intervention During the First 60 Days After Study Entry
Time Frame: Through 60 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: The Percentage of Patients Receiving Acute Therapeutic Intervention Beyond the First 60 Days After Study Entry
Time Frame: From 60 days through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: The Percentage of Platelet Counts ≥ 50,000/μl After Day 60 (If a Subject Receives an Acute Therapeutic Intervention, the Next Protocol-specified Platelet Count Will be Excluded From This Analysis, as it May be Influenced by the Intervention.)
Time Frame: From 60 days through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: The Percentage of Platelet Counts ≥ 150,000/μl After Day 60 (If a Subject Receives an Acute Therapeutic Intervention, the Next Protocol-specified Platelet Count Will be Excluded From This Analysis, as it May be Influenced by the Intervention.)
Time Frame: From 60 days through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: The Percentage of Patients Undergoing Splenectomy
Time Frame: Through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Change in the Quality of Life From Randomization to Weeks 4, 8 and End of Study, Determined Using the SF-36 Health Survey
Time Frame: Weeks 4, 8, and 52 after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: The Incidence and Severity of Bleeding as Defined by a Customized Bleeding Score
Time Frame: Through 365 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: The Percentage of Patients Not Completing Study Therapy
Time Frame: 49 days after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: The Percentage of Patients With Severe Adverse Events Attributable to Steroid Therapy
Time Frame: Through 1 year after study entry
Population: Due to the same sample size at the time that the study was terminated, this endpoint was not analyzed.
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | High Dose Pulse Dexamethasone | Standard Prednisone Therapy
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/3
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Pulse Dexamethasone (N=5) | Standard Prednisone Therapy (N=3)
Adverse drug reaction (General disorders) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Occult blood (Investigations) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose Pulse Dexamethasone (N=5) | Standard Prednisone Therapy (N=3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abnormal weight gain (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Anaemia vitamin B12 deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 5 (8) | 2 (2)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Application site bleeding (General disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (3) | 0 (0)
Chest pain (General disorders) | 3 (4) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (3)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Face oedema (General disorders) | 1 (2) | 1 (2)
Fat tissue increased (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 5 (8) | 3 (3)
Feeling jittery (General disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (6) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 4 (7) | 3 (3)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 5 (10) | 2 (4)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (4)
Libido decreased (Psychiatric disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Male sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 1 (4) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 3 (5) | 2 (2)
Mouth haemorrhage (Gastrointestinal disorders) | 2 (3) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucosal haemorrhage (General disorders) | 1 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Nail discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Nightmare (Psychiatric disorders) | 2 (2) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Occult blood (Investigations) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Oil acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onycholysis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (5) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Poor quality sleep (Nervous system disorders) | 2 (3) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 4 (4) | 2 (3)
Scleral haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 4 (5) | 2 (3)
Tremor (Nervous system disorders) | 1 (1) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Viral upper respiratory tract (Infections and infestations) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 5 (6) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Weight fluctuation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Compensatory sweating (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Menstrual cycle management (Surgical and medical procedures) | 1 (1) | 0 (0)
Skin discomfort (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No